CLINICAL TRIAL: NCT01731158
Title: A Prospective, Open-label, Multicenter, Randomized Phase II Trial: Sequential Therapy With BEvacizumab, RAd001 (Everolimus) and Tyrosinekinase Inhibitors (TKI) in Metastatic Renal Cell Carcinoma (mRCC) (BERAT Study)
Brief Title: Sequential Therapy in Metastatic Renal Cell Carinoma
Acronym: BERAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Society for Anticancer Drug Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C-II-008; 2011-005939-78 (EudraCT Number)
Record Dates: First submitted 2012-09-28; First posted 2012-11-21 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Interferon alpha-2; Everolimus; Sorafenib; pazopanib; Sunitinib

ARMS (2):
- arm A (Other): sequential therapy with approved drugs
  Avastin in combination with Roferon-A (first-line), Afinitor (second-line) and a TKI (Sutent, Nexavar or Votrient) (third-line)
  Interventions: Drug: Avastin in combination with Roferon-A; Drug: Afinitor; Drug: TKI: Sutent, Nexavar or Votrient
- arm B (Other): sequential therapy with approved drugs
  Avastin in combination with Roferon-A (first-line), a TKI (Sutent, Nexavar or Votrient) (second-line) and Afinitor (third-line)
  Interventions: Drug: Avastin in combination with Roferon-A; Drug: Afinitor; Drug: TKI: Sutent, Nexavar or Votrient

INTERVENTIONS:
Drug: Avastin in combination with Roferon-A
  Other Names: Bevacizumab in combination with Interfereon-alfa
Drug: Afinitor
  Other Names: Everolimus
Drug: TKI: Sutent, Nexavar or Votrient — TKI
  Other Names: Sunitinib, Sorafenib or Pazopanib

SUMMARY:
Sequential therapy with BEvacizumab, RAd001 (everolimus) and Tyrosinekinase inhibitors (TKI) in metastatic renal cell carcinoma (mRCC)

DETAILED DESCRIPTION:
This will be a prospective, open label, randomized multicenter phase-II study to evaluate progression free survival (PFS) in 2nd line treatment in patients with locally advanced or metastatic clear-cell renal cell cancer (cc-RCC) receiving everolimus (arm A) in comparison to a tyrosine-kinase inhibitor (TKI) (arm B). Following 2nd line treatment, patients will be switched to a TKI in arm A and everolimus in arm B. All patients will receive bevacizumab as standardized first-line treatment.

Another key element of the study is the analysis of predictive biomarkers, which will be performed in serum and tumor tissue, respectively. Serum samples will be collected at prespecified timepoints throughout the study and analysed by SELDI-TOF-MS and DIGE. Candidate proteins are thought to predict therapeutic outcome and candidates are subject for target validation by Western Blot or ELISA. In addition, formalin-fixed paraffin-embedded (FFPE) tumor tissue will be collected prospectively and analysed for micro RNA (miRNA). Candidate miRNAs that predict therapeutic outcome will be validated by quantitative RT-PCR. Furthermore, circulating tumor cells (CTCs) will be generated from blood drawings during routine visits. The primary objective is to correlate the marker profile defined from the FFPE tissue with the profile obtained from CTCs in order to validate expression based markers ant their change during different treatment lines.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Documented progressive disease prior to study inclusion.
* Adult males and females: ≥ 18 years of age.
* Metastatic or locally advanced RCC, not amendable to surgery with curative intention.
* ECOG performance status 0-1.
* Patients with measurable disease (at least one uni-dimensionally measurable target lesion by CT-scan or MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) If prior palliative radiotherapy to metastatic lesions: ≥ 1 measurable lesion that has not been irradiated. Patients with bone lesions as the only measurable lesion are eligible, provided that lesions consist of soft tissue, which is assessed via CT or MRI.
* Prior radiotherapy and surgery are allowed if completed 4 weeks (for minor surgery 2 weeks) prior to start of treatment and patient recovered from toxic effects.
* Modified MSKCC risk (according to Heng): good or intermediate.
* White blood cell count (WBC) ≥ 4x10*9/L with neutrophils ≥ 1.5 x 10*9/L, platelet count ≥ 100x10*9/L, hemoglobin ≥ 9 g/dL.
* Total bilirubin ≤ 2 x upper limit of normal.
* AST and ALT ≤ 2.5 x upper limit of normal, or ≤ 5 x upper limit of normal in case of liver metastases.
* Serum creatinine ≤ 2 x upper limit of normal or calculated creatinine clearance >30 ml/min.
* International Normalized Ratio (INR) ≤1.5 except for patients on stable anticoagulant therapy. Activated partial thromboplastin time (aPTT) ≤1.5 times upper limit of normal (ULN) or greater than the lower limit of the therapeutic range. Note: The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks at the treatment start.
* Adequate cardiac function (left ventricular ejection fraction ≥50% as assessed by ECHO)

Exclusion Criteria:

* Any investigational drug within the 30 days before inclusion.
* Known or suspected allergy or hypersensitivity reaction to any of the components of study treatments or their excipients.
* Pregnancy (absence to be confirmed by beta-hCG test) or lactation period.
* Men or women of child-bearing potential who are sexually active and unwilling to use a highly effective method of contraception (Pearl index < 1%) during the trial. Oral contraceptives are acceptable if a barrier method is applied in conjunction.
* Clinically symptomatic brain or meningeal metastasis (known or suspected), unless completion of local therapy for at least 3 months with discontinuation of steroids prior to start of treatment.
* Cardiac arrhythmias requiring anti-arrhythmics (excluding beta blockers, digoxin or digitoxin).
* History of any of the following cardiac events within the past 6 months:

  1. myocardial infarction (including severe/unstable angina),
  2. coronary/peripheral artery bypass graft,
  3. congestive heart failure (CHF) (NYHA Class III, or IV),
  4. cerebrovascular accident,
  5. transient ischemic attack,
  6. pulmonary embolism, abdominal or tracheo-oesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess
* Hemorrhage ≥ grade 3 or clinically significant hemoptysis within the past 4 weeks
* Uncontrolled severe hypertension (failure of diastolic blood pressure to fall below 90 mm Hg despite the use of ≥ 3 anti-hypertensive drugs).
* History of relevant pulmonary hypertension or interstitial lung disease or severely impaired lung function.
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease or chronic diarrhea.
* Previous malignancy (other than renal cell cancer) in the last 3 years, except basal cell cancer of the skin, pre-invasive cancer of the cervix, T1a prostate carcinoma or superficial bladder tumor [Ta, Tis and T1].
* History of organ allograft.
* Significant disease which, in the investigator's opinion would exclude the patient from the study.
* Medication that is known to interfere with any of the agents applied in the trial.
* Patients with a serious non-healing wound, ulcer or bone fracture.
* Patients with a history of seizure(s) not controlled with standard medical therapy.
* Patients receiving chronic systemic treatment with corticosteroids (dose of > 20 mg/day methylprednisone equivalent) or another immune-suppressive agent. Inhaled and topical steroids are acceptable.
* Legal incapacity or limited legal capacity.
* Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent.
* Significant vascular disease (e.g. aortic aneurysm, aortic dissection), or symptomatic peripheral vascular disease.
* Evidence or history of recurrent thromboembolism (>1 episode of deep venous thrombosis/peripheral embolism ≥ CTCAE Grade 3) during the past 2 years, bleeding diathesis or coagulopathy.
* Poorly controlled diabetes as defined by fasting serum glucose > 2.0 x ULN.
* Active (acute or chronic) or uncontrolled infection of bacterial, mycotic or viral genesis.
* Liver disease such as chronic active hepatitis or chronic persistent hepatitis.
* Patients with a known history of HIV seropositivity.
* QT prolongation (QTc > 450 msec).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
PFS rate of 2nd line treatment at 6 months after randomisation | 6 months after randomisation
  PFS rate

SECONDARY OUTCOMES:
PFS for 2nd line treatment | after completion of second-line treatment (expected median treatment 1st and 2nd line: 16 months)
  PFS
PFS for each treatment given | after completion of each treatment line (expected median treatment duration 1st line: 11 months, 2nd line: 5 months, 3rd line: 6 months)
  PFS
Overall Survival | after death of patient
  OS
number and severity (CTCAE 4.0) adverse events | continuously throughout trial
  AE
changes in quality of life throughout the Trial using FKSI questionnaires | continuously throughout trial (baseline, week 5, week 11, every 12 weeks, end of treatment for all treatment lines via FKSI-10 questionnaire)
  quality of life
ORR for each treatment given | after completion of each treatment line (expected median treatment duration 1st line: 11 months, 2nd line: 5 months, 3rd line: 6 months)
  ORR

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Grünwald, MD, Study Chair — University Hospital Hannover, Germany
Locations (13):
- Germany (13):
  - Charité Berlin, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Dresden, Dresden
  - University Hospital Düsseldorf, Düsseldorf
  - Waldkrankenhaus St. Marien, Erlangen
  - University Hospital Essen, Essen
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Göttingen, Göttingen
  - Oncological Practice Hannover, Hanover
  - University Hospital Hannover, Hanover
  - University Hospital Magdeburg, Magdeburg
  - University Hospital Tübingen, Tübingen

REFERENCES:
- [Derived] Nel I, Gauler TC, Bublitz K, Lazaridis L, Goergens A, Giebel B, Schuler M, Hoffmann AC. Circulating Tumor Cell Composition in Renal Cell Carcinoma. PLoS One. 2016 Apr 21;11(4):e0153018. doi: 10.1371/journal.pone.0153018. eCollection 2016. PMID 27101285